CLINICAL TRIAL: NCT00110656
Title: A Retrospective Follow Up Study to Evaluate the Status of Subjects That Discontinued Participation in a Qualifying Amgen Sponsored AMG 073 Study Due to Kidney Transplantation
Brief Title: Study To Evaluate the Status of Subjects That Discontinued Participation in a Qualifying Amgen Sponsored AMG 073 Study Due to Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20030219
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplant
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: None Retained — Retrospective data collected.

GROUPS / COHORTS (1):
- Kidney Transplant: All patients entered into the study will have received a kidney transplant.
  Interventions: Other: Observations

INTERVENTIONS:
Other: Observations — This is a non-interventional study- only observational.

SUMMARY:
The purpose of this study is to collect local laboratory data on immunoreactive parathyroid hormone (iPTH), calcium and phosphorus levels and estimated glomerular filtration rate (GFR) at approximately 1 week, 1 month, 3 months, 6 months and 12 months after the kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

- Patients who withdrew from one of the qualifying studies (i.e. patient previously took part in an Amgen study investigating the drug AMG 073 and its effects on secondary hyperparathyroidism [HPT]; in particular parathyroid hormone [PTH], calcium and phosphorus levels in blood associated with kidney failure) due to kidney transplantation.

Exclusion Criteria:

- Patient has any kind of disorder that compromises the ability of the subject to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Secondary HPT and ESRD who previously qualified for Amgen AM 073 studies but were withdrawn due to kidney transplant.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2004-03; Primary Completion 2004-09 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
PTH Values | 12 months post kidney translplant

SECONDARY OUTCOMES:
Calcium and Phosphorus | 12 months post kidney transplant

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com